CLINICAL TRIAL: NCT07271368
Title: AN EXTERNAL NEGATIVE PRESSURE USE DURING THE LISA PROCEDURE. A FEASIBILITY STUDY
Brief Title: EXTERNAL NEGATIVE PRESSURE DURING LISA
Acronym: ENCP LISA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Ján Hlivák, Principal investigator, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117/25 S-IV AP
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Neonatology
Keywords: LISA, negative pressure, neonatology, preterm, surfactant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Infants will remain on CPAP (6-8 cm H₂O) or HFNC (8 L/min) with FiO₂ titrated to maintain SpO₂ ≥92%. LISA catheter will be introduced under direct laryngoscopic vision 1-2 cm below the vocal cords. Two fractional boluses of surfactant (Curosurf, 200 mg/kg) will be administered within 2 minutes during ECNP support using Hayek RTX via a well-fitted thoracoabdominal cuirass. ECNP will be maintained at -10 cmH₂O throughout administration and for 10 minutes after. FiO₂ will not be reduced until SpO₂ stabilizes ≥92% and FiO₂ is ≤0.25.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENCP LISA (Experimental): Infants will remain on CPAP (6-8 cm H₂O) or HFNC (8 L/min) with FiO₂ titrated to maintain SpO₂ ≥92%. LISA catheter will be introduced under direct laryngoscopic vision 1-2 cm below the vocal cords. Two fractional boluses of surfactant (Curosurf, 200 mg/kg) will be administered within 2 minutes during ECNP support using Hayek RTX via a well-fitted thoracoabdominal cuirass. ECNP will be maintained at -10 cmH₂O throughout administration and for 10 minutes after. FiO₂ will not be reduced until SpO₂ stabilizes ≥92% and FiO₂ is ≤0.25.
  Interventions: Procedure: ENCP

INTERVENTIONS:
Procedure: ENCP — Surfactant will be given in two doses within 2 minutes while continuous negative pressure is applied using the Hayek RTX thoracoabdominal cuirass. Negative pressure will be maintained during and for 10 minutes after administration.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, safety, and preliminary effectiveness of applying external continuous negative pressure (ECNP) during less invasive surfactant administration (LISA) in preterm infants with respiratory distress syndrome (RDS). It will also assess whether ECNP can improve surfactant distribution and reduce procedural complications. The main questions it aims to answer are:

Does ECNP during LISA improve surfactant distribution and oxygenation in preterm infants with RDS?

Does ECNP reduce the occurrence of complications such as desaturation, bradycardia, or apnea during the procedure?

Does ECNP reduce the need for repeated surfactant administration?

Researchers will evaluate ECNP combined with LISA in preterm infants on HFNC or CPAP to see if it improves outcomes compared to standard methods.

Participants will:

Receive LISA with ECNP support via a soft thoracoabdominal cuirass

Be monitored for procedural complications like desaturation, bradycardia, or apnea

Have their oxygenation levels, surfactant distribution, and need for repeated surfactant doses assessed

Primary Outcome:

The procedure will be considered safe if no more than 20% of participants experience serious adverse events, such as apnea requiring positive pressure ventilation or persistent desaturation.

Secondary Outcomes:

Completion of LISA without interruption due to complications

Reduction of FiO₂ to ≤0.25 within 3 hours post-surfactant administration

Avoidance of repeated surfactant doses via the INSURE method

DETAILED DESCRIPTION:
This pilot study evaluates the feasibility, safety, and preliminary effectiveness of applying external continuous negative pressure (ECNP) during less invasive surfactant administration (LISA) in preterm infants with respiratory distress syndrome (RDS) supported by non-invasive respiratory support. ECNP, delivered via a modern negative-pressure ventilation device and a soft thoracoabdominal cuirass, generates a sustained sub-atmospheric pressure around the chest wall. This mode of support is intended to facilitate spontaneous breathing, promote more homogeneous lung inflation, and potentially enhance the distribution of intratracheally delivered surfactant.

LISA using thin catheters is a widely adopted method for surfactant administration in spontaneously breathing neonates receiving CPAP or HFNC. Although effective, the procedure is frequently complicated by transient hypoxemia, bradycardia, apnea, and surfactant reflux, occasionally requiring temporary interruption or conversion to more invasive therapy. These complications may impair surfactant delivery, contribute to uneven lung aeration, and lead to the need for repeated dosing. To date, the integration of continuous negative-pressure support during LISA has not been evaluated in clinical practice.

In this single-arm feasibility study, ECNP will be initiated shortly before and maintained throughout the LISA procedure. The study will assess whether negative-pressure support stabilizes spontaneous ventilation, improves oxygenation, and facilitates more uniform surfactant distribution during administration. Safety will be evaluated based on the occurrence of serious procedure-related events requiring interruption, such as significant desaturation, bradycardia, or apnea requiring positive-pressure ventilation. Effectiveness will be explored through measures of post-procedure oxygenation stability, need for repeat surfactant dosing, and indicators of adequate surfactant distribution (e.g., imaging assessments when clinically indicated).

This exploratory study is designed to inform the potential utility of ECNP as an adjunct during LISA and to determine whether a larger controlled trial is warranted. The protocol focuses on documenting feasibility (ability to complete LISA under ECNP), characterizing physiologic responses, and capturing any adverse events specifically associated with ECNP use in this population

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≥ 32 weeks of gestational age
* FiO₂ > 0.30 for more than 30 minutes on CPAP (6 - 8 cm H₂O) or HFNC (8 l/min)
* Increased work of breathing despite FiO₂ < 0.30
* Birth weight > 800 g
* X-ray confirmed RDS
* Availability of all required devices and appropriately fitting cuirass

Exclusion Criteria:

* Requirement for endotracheal intubation or mechanical ventilation prior to surfactant administration
* Major congenital anomalies (cardiac, pulmonary, chromosomal)
* Known or suspected neuromuscular or metabolic disorders
* Lack or withdrawal of informed parental consent

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety of the procedure | 15 minutes
  No more than 20% of neonates experience serious adverse events requiring procedural interruption.
  Serious adverse events:
  * apnea necessitating positive pressure ventilation (PPV) or intubation
  * persistent desaturation (SpO₂ < 80%) unresponsive to increased FiO₂
  * prolonged bradycardia (heart rate < 100 bpm) requiring interruption of the procedure
  * any other adverse event or treatment failure leading to the need for a repeated surfactant administration.

SECONDARY OUTCOMES:
Completion of the LISA procedure without interruption | 3 hours
  Completion of the LISA procedure without interruption due to desaturation, bradycardia, or apnea, and reduction of FiO₂ to ≤0.25 within 3 hours after surfactant administration.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deep A, De Munter C, Desai A. Negative pressure ventilation in pediatric critical care setting. Indian J Pediatr. 2007 May;74(5):483-8. doi: 10.1007/s12098-007-0082-2. PMID 17526961
- [Background] Kribs A, Roll C, Gopel W, Wieg C, Groneck P, Laux R, Teig N, Hoehn T, Bohm W, Welzing L, Vochem M, Hoppenz M, Buhrer C, Mehler K, Stutzer H, Franklin J, Stohr A, Herting E, Roth B; NINSAPP Trial Investigators. Nonintubated Surfactant Application vs Conventional Therapy in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):723-30. doi: 10.1001/jamapediatrics.2015.0504. PMID 26053341
- [Background] Aldana-Aguirre JC, Pinto M, Featherstone RM, Kumar M. Less invasive surfactant administration versus intubation for surfactant delivery in preterm infants with respiratory distress syndrome: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F17-F23. doi: 10.1136/archdischild-2015-310299. Epub 2016 Nov 15. PMID 27852668
- [Background] Dargaville PA, Aiyappan A, Cornelius A, Williams C, De Paoli AG. Preliminary evaluation of a new technique of minimally invasive surfactant therapy. Arch Dis Child Fetal Neonatal Ed. 2011 Jul;96(4):F243-8. doi: 10.1136/adc.2010.192518. Epub 2010 Oct 21. PMID 20971722
- [Background] Roberts CT, Halibullah I, Bhatia R, Green EA, Kamlin COF, Davis PG, Manley BJ. Outcomes after Introduction of Minimally Invasive Surfactant Therapy in Two Australian Tertiary Neonatal Units. J Pediatr. 2021 Feb;229:141-146. doi: 10.1016/j.jpeds.2020.10.025. Epub 2020 Oct 14. PMID 33068569
- [Background] Dargaville PA, Ali SKM, Jackson HD, Williams C, De Paoli AG. Impact of Minimally Invasive Surfactant Therapy in Preterm Infants at 29-32 Weeks Gestation. Neonatology. 2018;113(1):7-14. doi: 10.1159/000480066. Epub 2017 Sep 19. PMID 28922658
- [Background] Kurepa D, Perveen S, Lipener Y, Kakkilaya V. The use of less invasive surfactant administration (LISA) in the United States with review of the literature. J Perinatol. 2019 Mar;39(3):426-432. doi: 10.1038/s41372-018-0302-9. Epub 2019 Jan 11. PMID 30635595
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Mohammadizadeh M, Ardestani AG, Sadeghnia AR. Early administration of surfactant via a thin intratracheal catheter in preterm infants with respiratory distress syndrome: Feasibility and outcome. J Res Pharm Pract. 2015 Jan-Mar;4(1):31-6. doi: 10.4103/2279-042X.150053. PMID 25710048
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476